CLINICAL TRIAL: NCT05802056
Title: COordinated Nivolumab and IntraperiToneal IL-2 for Gastric CanceR With PeritOneaL Metastasis (CONTROL) Phase 1b Pilot Study
Brief Title: Aldesleukin With Nivolumab and Standard Chemotherapy for Treatment of Gastric Cancer With Peritoneal Metastasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC220404; NCI-2023-02250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC220404 (Other: Mayo Clinic); 22-009956 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage IV Gastric Cancer AJCC v8; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Metastatic Gastric Carcinoma; Metastatic Malignant Neoplasm in the Peritoneum
MeSH Terms: conditions — Stomach Neoplasms | interventions — aldesleukin; Biopsy; Specimen Handling; Laparoscopy; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Nivolumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (aldesleukin, nivolumab, chemotherapy) (Experimental): Patients receive aldesleukin IP over at least 40 minutes on days 1 and 8 of each cycle. Patients also receive standard of care nivolumab IV over 30 minutes on day 1, leucovorin calcium IV over 2 hours on day 1, oxaliplatin IV over 2 hours on day 1, and flurouracil IV continuously over 46 hours on days 1-3 for each cycle. Cycles repeat every 14 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo diagnostic laparoscopy with biopsy, PET/CT or PET/MRI, and collection of blood and tissue samples throughout the trial.
  Interventions: Biological: Aldesleukin; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Diagnostic Laparoscopy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Oxaliplatin; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Aldesleukin — Given IP
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography; Computerized axial tomography (procedure); Computerized Tomography (CT) scan
Procedure: Diagnostic Laparoscopy — Undergo diagnostic laparoscopy
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); MRIs; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo; ABP 206; BCD-263; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT; Positron emission tomography (procedure)

SUMMARY:
This phase Ib trial test effects of aldesleukin in combination with nivolumab and standard chemotherapy in treating patients with gastric cancer that has spread to the tissue lining of the abdomen (peritoneal metastasis). Aldesleukin is similar to a protein that naturally exists in the body that stimulates the immune system to fight infections. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as leucovorin calcium, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving aldesleukin in combination with nivolumab and standard chemotherapy may work better in treating patients with gastric cancer with peritoneal metastasis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the reduction in the peritoneal carcinomatosis index (PCI) after completion of the study treatment.

SECONDARY OBJECTIVES:

I. Evaluate histological response of the peritoneal metastasis to study treatment using the peritoneal regression grading score (PRGS).

II. Assess overall survival (OS). III. Assess progression-free survival (PFS). IV. Assess safety and tolerability of the study regimen.

TERTIARY AND CORRELATIVE RESEARCH OBJECTIVES:

I. Assess the number and percentage of patients that successfully undergo complete cytoreductive surgery after treatment.

II. Evaluate for helper T cell, cytotoxic T cell, natural killer (NK) cells as well as T-reg cells in blood and peritoneal fluid.

III. Evaluate the neutrophilic, lymphocytic, and eosinophilic infiltration of tumor using a standardized classification.

OUTLINE:

Patients receive aldesleukin intraperitoneally (IP) over at least 40 minutes on days 1 and 8 of each cycle. Patients also receive standard of care nivolumab intravenously (IV) over 30 minutes on day 1, leucovorin calcium IV over 2 hours on day 1, oxaliplatin IV over 2 hours on day 1, and flurouracil IV continuously over 46 hours on days 1-3 for each cycle. Cycles repeat every 14 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo diagnostic laparoscopy with biopsy, positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI), and collection of blood and tissue samples throughout the trial.

After completion of study treatment, patients follow up at 30 days, 90 days then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Age >= 18 years
* PRE-REGISTRATION: Disease characteristics

  * Histological confirmation of adenocarcinoma of the stomach or gastroesophageal junction (GEJ)
  * Currently receiving first-line therapy with leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX) and nivolumab without evidence of disease progression OR planning to start first-line therapy with FOLFOX and nivolumab
* PRE-REGISTRATION: No radiographic or histological evidence of non-peritoneal metastasis
* PRE-REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* PRE-REGISTRATION: Willingness to provide mandatory blood specimens for correlative research
* PRE-REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research
* PRE-REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* REGISTRATION: Peritoneal Carcinomatosis Index (PCI) >= 1 and =< 24 obtained =< 30 days prior to registration
* REGISTRATION: Clinical, pathological, or radiographic evidence of peritoneal metastasis per PCI and Peritoneal Regression Grading Score (PRGS)
* REGISTRATION: Hemoglobin >= 8.0 g/dL (obtained =< 30 days prior to registration)
* REGISTRATION: Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 30 days prior to registration)
* REGISTRATION: Platelet count >= 75,000/mm^3 (obtained =< 30 days prior to registration)
* REGISTRATION: Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 30 days prior to registration)
* REGISTRATION: Alanine aminotransferase (ALT) AND aspartate transaminase (AST) =< 1.5 x ULN (obtained =< 30 days prior to registration)
* REGISTRATION: Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy, then INR or aPTT is within target range of therapy (obtained =< 30 days prior to registration)
* REGISTRATION: Calculated creatinine clearance >= 40 ml/min using the Cockcroft-Gault formula (obtained =< 30 days prior to registration)
* REGISTRATION: Negative pregnancy test done =< 8 days prior to registration, for persons of childbearing potential only
* REGISTRATION: Provide written informed consent
* REGISTRATION: Willingness to provide mandatory blood specimens for correlative research
* REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* PRE-REGISTRATION: Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* PRE-REGISTRATION: Any of the following prior therapies: IL-2 or chronic corticosteroids, or immunosuppressive agents

  * NOTE: Inhaled corticosteroids are allowed
* PRE-REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* PRE-REGISTRATION: Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* PRE-REGISTRATION: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
  * Autoimmune disease
* PRE-REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* PRE-REGISTRATION: Active second malignancy currently receiving systemic treatment =< 6 months prior to pre-registration
* PRE-REGISTRATION: History of myocardial infarction =< 6 months prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* REGISTRATION: Identification of non-peritoneal metastasis during laparoscopy
* REGISTRATION: Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* REGISTRATION: Any of the following therapies: prior immune checkpoint inhibitors, prior IL-2, or chronic corticosteroids or immunosuppressive agents

  * NOTE: Inhaled corticosteroids are allowed. One-time antiemetic dose is allowed
* REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* REGISTRATION: Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy
* REGISTRATION: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations (e.g., substance abuse) that would limit compliance with study requirements
  * Autoimmune disease requiring systemic treatment
  * Small bowel obstruction
* REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* REGISTRATION: History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* REGISTRATION: Small bowel obstruction < 15 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
Change of reduction in the peritoneal carcinomatosis index | About 90 days after last dose of aldesleukin (IL-2)
Incidence of adverse events | About 90 days after last dose of aldesleukin (IL-2)

SECONDARY OUTCOMES:
Histological response of the peritoneal metastasis | About 90 days after last dose of aldesleukin (IL-2)
  Will be assessed using the peritoneal regression grading score. Will be reported descriptively, including reporting of frequencies, percentages and 95% confidence intervals.
Progression free survival | From study entry to the first of either disease progression or death, assessed up to 3 years
  Summary statistics, including the median and other various timepoints will be reported as well as 95% confidence intervals.
Overall survival | From date of study entry to date of death or last follow up, assessed up to 3 years
  Summary statistics, including the median and other various timepoints will be reported as well as 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Travis E. Grotz, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials